CLINICAL TRIAL: NCT01797185
Title: Safety Study of SPARC1104
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLR_11_04
Record Dates: First submitted 2013-02-16; First posted 2013-02-22 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Spasticity
Keywords: spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SPARC1104 group 1 (Experimental)
  Interventions: Drug: SPARC1104 modified dose regimen I
- SPARC1104 group 2 (Experimental)
  Interventions: Drug: SPARC1104 modified dose regimen II
- SPARC1104 group 3 (Experimental)
  Interventions: Drug: SPARC1104 modified dose regimen III

INTERVENTIONS:
Drug: SPARC1104 modified dose regimen I — Subjects who exited study CLR_09_21
  Arms: SPARC1104 group 1
Drug: SPARC1104 modified dose regimen II — Subjects who received prior treatment regimen I
  Arms: SPARC1104 group 2
Drug: SPARC1104 modified dose regimen III — Subjects who received no prior treatment regimen
  Arms: SPARC1104 group 3

SUMMARY:
Open-label, safety study of SPARC1104 in subjects with spasticity due to multiple sclerosis

DETAILED DESCRIPTION:
Safety study of SPARC1104

ELIGIBILITY:
* Willingness to participate and give written informed consent
* Men and women ≥ 18 years of age
* Sexually active women who are of child bearing potential will practice an acceptable method of birth control for the duration of the trial as judged by the investigator. Examples of acceptable contraception are: condoms, foams, jellies, diaphragm, intrauterine device, oral or long-acting injected contraceptives, bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or having a partner who is incapable of initiating conception. The practice of contraception must have started at least 3 months prior to trial entry.
* If female, negative pregnancy test result at Screening
* Diagnosed with MS and a known history of spasticity
* Meet one of the following criteria o Subjects who completed the double-blind randomized withdrawal phase (Part 3) of trial CLR_09_21 with no major protocol violation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2013-04-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (51):
  - SPARC site 4, Gilbert, Arizona
  - SPARC Site 34, Phoenix, Arizona
  - SPARC Site 1, Tucson, Arizona
  - SPARC Site 30, Costa Mesa, California
  - SPARC Site 14, Newport Beach, California
  - SPARC Site 32, Basalt, Colorado
  - SPARC Site 5, Denver, Colorado
  - SPARC Site 7, Derby, Connecticut
  - SPARC site 47, Hartford, Connecticut
  - SPARC Site 8, New London, Connecticut
  - SPARC Site 50, Washington D.C., District of Columbia
  - SPARC Site 35, Maitland, Florida
  - SPARC Site 59, Miami, Florida
  - SPARC Site 6, Ormond Beach, Florida
  - SPARC Site 11, Port Charlotte, Florida
  - SPARC Site 13, Sarasota, Florida
  - SPARC Site 25, Sunrise, Florida
  - SPARC Site 55, Tampa, Florida
  - SPARC Site 33, Tampa, Florida
  - SPARC site 45, Lenexa, Kansas
  - SPARC Site 24, Overland Park, Kansas
  - SPARC Site 44, Louisville, Kentucky
  - SPARC site 36, Alexandria, Louisiana
  - SPARC Site 21, Baton Rouge, Louisiana
  - SPARC Site 61, New Orleans, Louisiana
  - SPARC Site 49, Baltimore, Maryland
  - SPARC Site 22, Fulton, Maryland
  - SPARC Site 29, Foxborough, Massachusetts
  - SPARC Site 17, Springfield, Massachusetts
  - SPARC Site 26, Clinton Township, Michigan
  - SPARC Site 54, Detroit, Michigan
  - SPARC Site 19, Golden Valley, Minnesota
  - SPARC Site 28, Flemington, New Jersey
  - SPARC Site 16, Albuquerque, New Mexico
  - SPARC Site 43, Rochester, New York
  - SPARC Site 52, White Plains, New York
  - SPARC site 39, Charlotte, North Carolina
  - SPARC Site 18, Greensboro, North Carolina
  - SPARC Site 2, Winston-Salem, North Carolina
  - SPARC Site 27, Centerville, Ohio
  - SPARC site 10, Eugene, Oregon
  - SPARC site 38, Springfield, Oregon
  - SPARC Site 57, Abington, Pennsylvania
  - SPARC Site 23, Old Point Station, South Carolina
  - SPARC Site 5, Austin, Texas
  - SPARC Site 60, Dallas, Texas
  - SPARC Site 37, Houston, Texas
  - SPARC Site 20, Tacoma, Washington
  - SPARC Site 62, Huntington, West Virginia
  - SPARC Site 58, Milwaukee, Wisconsin
  - SPARC Site 56, Waukesha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- SPARC1104 Group 1: Subjects who completed Part 3 of Study CLR_09_21 Dose: One or two capsules once daily
- SPARC1104 Group 2: Subjects who are on Dose regimen I of SPARC0921 at entry. Dose: One or two capsules once daily
- SPARC1104 Group 3: Subjects Entering the Trial with no Prior Treatment with SPARC0921 Dose: One or two capsules once daily
Period: Overall Study
Arm/Group | SPARC1104 Group 1 | SPARC1104 Group 2 | SPARC1104 Group 3
Started | 162 | 163 | 50
Completed | 134 | 125 | 38
Not Completed | 28 | 38 | 12
Not completed — Adverse Event | 5 | 15 | 6
Not completed — Withdrawal by Subject | 6 | 9 | 5
Not completed — Site terminated | 8 | 4 | 0
Not completed — Lost to Follow-up | 2 | 6 | 1
Not completed — Withdrawn per sponsor | 5 | 0 | 0
Not completed — Physician Decision | 1 | 3 | 0
Not completed — Protocol Violation | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- SPARC1104 Group 1: Subjects who completed Study CLR_09_21
- SPARC1104 Group 2: Subjects who are on Dose regimen I of SPARC0921 at entry
- SPARC1104 Group 3: Subjects Entering the Trial with no Prior Treatment with SPARC0921
- Total: Total of all reporting groups
Arm/Group | SPARC1104 Group 1 | SPARC1104 Group 2 | SPARC1104 Group 3 | Total
Number analyzed (Participants) | 162 | 163 | 50 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (9.56) | 52.9 (9.77) | 51.3 (11.55) | 52.2 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 116 | 29 | 264
  Male | 43 | 47 | 21 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 3 | 15
  Not Hispanic or Latino | 155 | 158 | 47 | 360
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 28 | 19 | 5 | 52
  White | 132 | 139 | 44 | 315
  More than one race | 1 | 4 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Time Frame: 52 weeks
Population: Safety population: Subject who received at least one dose of study treatment
Measure: Number; unit: Count of participants
Arm/Group | SPARC1104 Group 1 | SPARC1104 Group 2 | SPARC1104 Group 3
Number analyzed (Participants) | 162 | 163 | 50
Count of participants | 129 | 150 | 44

ADVERSE EVENTS:
Time Frame: Week 26
Arm/Group | SPARC1104 Group 1 | SPARC1104 Group 2 | SPARC1104 Group 3
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/163 | 0/50
Serious Adverse Events (participants affected / at risk) | 30/162 | 40/163 | 6/50
Other Adverse Events (participants affected / at risk) | 129/162 | 150/163 | 44/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPARC1104 Group 1 (N=162) | SPARC1104 Group 2 (N=163) | SPARC1104 Group 3 (N=50)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Acquired oesophageal web (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 4 | 5 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0
Partial seizures (Nervous system disorders) | 1 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0
Complex partial seizures (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 3 | 5 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 0 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPARC1104 Group 1 (N=162) | SPARC1104 Group 2 (N=163) | SPARC1104 Group 3 (N=50)
Headache (Nervous system disorders) | 26 | 31 | 11
Multiple sclerosis relapse (Nervous system disorders) | 29 | 30 | 7
Muscle spasticity (Nervous system disorders) | 24 | 32 | 9
Urinary tract infection (Nervous system disorders) | 32 | 21 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 35 | 4
Nausea (Gastrointestinal disorders) | 19 | 24 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 26 | 4
Fatigue (General disorders) | 16 | 25 | 5
Dizziness (Nervous system disorders) | 11 | 22 | 11
Fall (Injury, poisoning and procedural complications) | 20 | 22 | 2
Nasopharyngitis (Infections and infestations) | 13 | 23 | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 14 | 23 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 20 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 19 | 4
Diarrhoea (Gastrointestinal disorders) | 16 | 14 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 22 | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 7 | 16 | 4
Insomnia (Psychiatric disorders) | 10 | 15 | 2
Upper respiratory tract infection (Infections and infestations) | 11 | 11 | 2
Sinusitis (Infections and infestations) | 10 | 12 | 0
Hypoaesthesia (Nervous system disorders) | 7 | 9 | 5
Vomiting (Gastrointestinal disorders) | 12 | 7 | 2
Asthenia (General disorders) | 9 | 9 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 10 | 1
Oedema peripheral (General disorders) | 8 | 11 | 1
Depression (Psychiatric disorders) | 8 | 8 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 9 | 10 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2015-12-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT01797185/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT01797185/SAP_001.pdf